CLINICAL TRIAL: NCT06697834
Title: Assessment of Pain in Plantar Fasciitis Managed by Histotripsy
Acronym: HISTO-APS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01296-39
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Fasciitis, Plantar; Aponeurosis Contusion
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with plantar fasciitis (Experimental)
  Interventions: Procedure: Histotripsy ultrasound session; Other: VAS questionnaire; Other: AOFAS questionnaire

INTERVENTIONS:
Procedure: Histotripsy ultrasound session — The study will be performed with the MINDRAY DP-10 ultrasound device equipped with a linear probe and histotripsy functionality.
Other: VAS questionnaire — Pain assessment with the EVA questionnaire
Other: AOFAS questionnaire — AOFAS questionnaire at visit 1 and visit 4 (75 days after the first visit).

SUMMARY:
Plantar fasciitis or plantar fasciitis is the most commonly reported cause of pain under the heel. Its prevalence varies from 3.6 to 7% in the general population. It is a painful condition of the foot that corresponds to an inflammation of the plantar fascia.

At present, histotripsy in the field of orthopedics is very little used. The concept of therapeutic ultrasound intended for the treatment of plantar fasciitis by fascial section was developed in the United States but no study evaluating its effects on pain is available.

There is no equivalent study on histotripsy in the pathology of chronic plantar fasciitis or fasciitis. In this study, histotripsy will be performed using a conventional serial ultrasound system with this focused energy function.

The research hypothesis is that histotripsy treatment may be an alternative to pain management in patients with plantar fasciitis who have failed conventional treatments.

The main objective of this study is to evaluate the evolution of the pain felt by patients with plantar fasciitis resistant to conventional medical treatment, one month after two ultrasound histotripsy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 years minimum
* Patient with plantar fasciitis evolving for at least 6 months
* Patients with radiology and MRI of the foot less than 3 months old
* Visual analogue pain scale greater than 5 at inclusion
* Patient in whom conventional medical treatment has failed by the combination of radial shock waves, plantar orthoses, and corticosteroid infiltration that has not provided relief.
* Patient affiliated with or beneficiary of a social security scheme.
* Patient who has been informed and has given his/her free, informed and written consent.

Exclusion Criteria:

* Minor patient
* Major retraction of the triceps surae on the MAESTRO oblique board test: sequelae of bone trauma to the hindfoot and ankle.
* Inflammatory rheumatological diseases
* Fibromyalgia
* Patients in whom a specific underlying organic pathology (inflammatory, infectious, neoplastic, etc.) has been identified.
* Psychiatric disorders
* Patient participating in another research study.
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman.
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
the percentage of change in pain (VAS 0-10) | 1 month and a half
  the percentage of change in pain (VAS 0-10) felt 1 month after two ultrasound histotripsy sessions (visit 4) compared to the baseline value (visit 1).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de Domont, Domont, France